CLINICAL TRIAL: NCT05295966
Title: Effects of Multisensory Physical Exercises in People With Moderate Cognitive Impairment or Mild Dementia
Brief Title: Multisensory Physical Exercises in People With Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Miguel Fernández del Olmo, Proffessor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V1058
Record Dates: First submitted 2022-02-21; First posted 2022-03-25 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2022-03

CONDITIONS: Dementia
Keywords: Exercise; rehabilitation; sensory stimulation
MeSH Terms: conditions — Dementia; Motor Activity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Subjects in the intervention group will perform 20 sessions of multisensory training
  Interventions: Other: Cognitive therapy; Behavioral: Physiocognitive Integration
- Control Group (Active Comparator): Subjects in the Control Group will not perform 20 sessions of multisensory training and they will keep doing the current therapy
  Interventions: Other: Cognitive therapy

INTERVENTIONS:
Other: Cognitive therapy — Cognitive therapy
Behavioral: Physiocognitive Integration — Physiocognitive Integration
  Arms: Intervention Group

SUMMARY:
The main objective of the study is to evaluate the efficacy of a combined training program of physical exercise and multisensory stimulation (Physiocognitive Integration) in people with mild/moderate cognitive impairment.

DETAILED DESCRIPTION:
Alzheimer's disease and other dementias are the main cause of cognitive impairment, with a prevalence of 0.4% worldwide and 1.23 in Europe. The WHO estimates that the growth of people with cognitive impairment to some degree will increase in the coming years, exceeding 75 million people in the world in 2030, and 135 million in 2050. The prevention of cognitive deterioration is mainly based on the implementation of non-pharmacological therapies. Multisensory stimulation is a non-pharmacological therapy that has benefits in patients with cognitive impairment, producing an improvement in cognitive function.

Physical exercise is associated with a lower risk of onset of cognitive impairment and less cognitive impairment as well as a slower progression in people with mild cognitive impairment and in mild-stage dementias. In addition to the cognitive sphere, the positive effect of physical exercise in preventing falls has been widely studied.

The main objective of the study is to evaluate the efficacy of a combined training program of physical exercise and multisensory stimulation (Physiocognitive Integration) in people with mild/moderate cognitive impairment. In order to do this, a experimental group will perform 20 sessions of multisensory training in addition to their current therapy and a second, control group, only their current therapy. Before and after the time need to complete the 20 sessions, all subjects were perform a battery of motor and cognitive tasks.

ELIGIBILITY:
Inclusion Criteria:

* Absence of treatment with psychotropic drugs or stable dose of the same (without drug or dose modifications in the last four weeks).

In the case of subjects who are part of the intervention group, the following will also be inclusion criteria:

* Caregiver or family member who presents the appropriate skills for collaboration in the implementation of the exercises and in the management of the mobile application.
* Availability of the necessary time for the initial training in the handling of the devices, the development of the sessions and the communication with the researchers.

Exclusion Criteria:

* Insufficient physical condition for participation.
* Sensory deficits that make participation difficult.
* Unstable clinical situation.
* Unstable mental disorder or not adequately controlled with medication (depression, agitation, etc.).
* Presence of associated pathology that involves treatment with drugs that alter cognitive abilities or interfere with the user's participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Speed of Gait at preferred pace | baseline
  Variables: Speed (m/s)
Speed of Gait at preferred pace | at week 8
  Variables: Speed (m/s)
Cadence of Gait at preferred pace | baseline
  Variables: cadence (steps/min)
Cadence of Gait at preferred pace | at week 8
  Variables: cadence (steps/min)
Step Length of Gait at preferred pace | baseline
  Variables: Step Length (m)
Step Length of Gait at preferred pace | at week 8
  Variables: Step Length (m)
Speed during Dual task gait | baseline
  Variables: Speed (m/s)
Speed during Dual task gait | at week 8
  Variables: Speed (m/s)
Cadence during Dual task gait | Baseline
  Variables: cadence (steps/min)
Cadence during Dual task gait | at week 8
  Variables: cadence (steps/min)
Step Length during Dual task gait | Baseline
  Variables: Step Length (m)
Step Length during Dual task gait | at week 8
  Variables: Step Length (m)
Time up & go test | baseline
  Variables: time (seconds)
Time up & go test | at week 8
  Variables: time (seconds)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Rey Juan Carlos, Fuenlabrada, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided